CLINICAL TRIAL: NCT03535870
Title: A Randomized, Parallel-Group, Placebo-Controlled, Clinical Endpoint Bioequivalence Study of Generic Fluticasone Propionate 100 μg and Salmeterol Xinafoate 50 μg Inhalation Powder Compared With Advair Diskus® 100/50 in Subjects With Asthma
Brief Title: Clinical Endpoint Bioequivalence Study of Fluticasone Propionate & Salmeterol Xinafoate (100μg/50μg)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West-Ward Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLSA-P100/50-PVCL-2
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluticasone propionate/salmeterol (Experimental): fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) twice a day by inhalation throughout the study
  Interventions: Drug: Fluticasone propionate/salmeterol
- Advair Diskus, 100 Mcg-50 Mcg Inhalation Powder (Active Comparator): Advair Diskus (fluticasone propionate and salmeterol xinafoate) twice a day by inhalation throughout the study
  Interventions: Drug: Advair Diskus, 100 Mcg-50 Mcg Inhalation Powder
- Placebo (Placebo Comparator): placebo inhaled powder twice a day by inhalation throughout the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered via the LOMI inhaler device
  Arms: Fluticasone propionate/salmeterol
Drug: Advair Diskus, 100 Mcg-50 Mcg Inhalation Powder — Advair (Fixed dose combination of fluticasone propionate and salmeterol xinafoate administered via the Diskus inhaler device)
  Arms: Advair Diskus, 100 Mcg-50 Mcg Inhalation Powder
Drug: Placebo — placebo dry powder administered via the LOMI inhaler device
  Arms: Placebo

SUMMARY:
A Randomized, Parallel-Group, Placebo-Controlled, Clinical Endpoint Bioequivalence Study of Generic Fluticasone Propionate 100 μg and Salmeterol Xinafoate 50 μg Inhalation Powder Compared with Advair Diskus® 100/50 in Subjects with Asthma

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical bioequivalence of generic fluticasone propionate 100 μg and salmeterol xinafoate 50 μg inhalation powder (test) to Advair Diskus ("Advair") 100/50 (reference) for the treatment of asthma.

The secondary objectives of the study are:

* To demonstrate statistical superiority of generic fluticasone propionate 100 μg and salmeterol xinafoate 50 μg inhalation powder to placebo.
* To demonstrate statistical superiority of Advair 100/50 to placebo.
* To investigate the safety and tolerability of fluticasone propionate 100 μg and salmeterol xinafoate 50 μg inhalation powder compared with Advair 100/50 in the target population

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects must be 12 years of age or older.
2. Females must not be of childbearing potential or if of childbearing potential, must commit to consistent use of a form of birth control which is medically effective, in the judgment of the investigator.
3. Be able to provide written informed consent or, in the case of adolescents, informed assent in addition to an informed consent form (ICF) signed by the adolescent's parent(s) or legal guardian(s).
4. Be current non-smokers and also may not have used tobacco products (e.g., cigarettes, e-cigarettes, cigars, pipe tobacco) within the year prior to Visit 1, and have 10 years or less (10 pack-years for cigarettes) of historical use.
5. Have persistent asthma, as defined by the National Asthma Education and Prevention Program, for at least 12 weeks before Visit 1.
6. FEV1 at Visit 1 (screening) and Visit 2 (randomization) of: ≥40% and ≤85% predicted normal value (for age ≥18 years), or ≥65% and ≤85% predicted normal value (for ages 12 to 17 years)
7. Demonstrate ≥15% reversibility of FEV1 between 10 and 30 minutes following 360 μg of albuterol inhalation. This may be demonstrated at the Screening Visit or anytime in the period leading up to Visit 2 (randomization).
8. Be able to discontinue controller asthma medication (including LTM, inhaled corticosteroids [ICS] and long-acting β-agonists (LABAs]) during the Run-in Period and Treatment Period.
9. Be able to replace current short-acting β-agonists (SABAs) with the study-supplied albuterol (or equivalent) rescue medication inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for a least 6 hours before lung function assessments during study visits).
10. Must not have been treated (for any reason) with oral or parenteral corticosteroids for at least 1 month before Visit 1 and must not have used oral SABAs (not inhaled) for at least 12 hours before Visit 1 and for the remainder of the study. Use of oral/parenteral corticosteroids and oral SABAs is prohibited after Visit 1.
11. Subjects may continue using short-acting forms of theophylline (withheld at least 12 hours before study visits), twice daily controlled-release forms of theophylline (withheld at least 24 hours before study visits), and once daily controlled-release forms of theophylline (withheld at least 36 hours before study visits). Subjects must be judged by the investigator as able to withhold these medications for the specified minimum time intervals before each site visit.
12. Be able to answer questions regarding asthma status and be able to document device usage and asthma status on a twice daily basis.
13. Demonstrate proper use of MDI and dry-powder inhaler devices.

Exclusion Criteria:

1. Have a FEV1 reversibility of <15% at Visit 1.
2. Are unable to discontinue ICS, LABA, or LTM.
3. Have a history of life-threatening asthma, defined as an asthma episode (at any time in the past) associated with any of the following: respiratory arrest or intubation, hypercapnia, hypoxic seizures, or syncopal episode.
4. Have a hospitalization within the year prior to Screening due to an asthma exacerbation.
5. Have exercise-induced asthma as the only asthma-related diagnosis that does not require daily asthma control medicine.
6. Have evidence or history of congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia.
7. Have evidence or history of any disease (hematologic, hepatic, neurologic, psychiatric, renal, or other) that in the opinion of the investigator, would put the subject at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
8. Have any other relevant pulmonary disease except for asthma, including but not limited to chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, bronchiectasis, chronic bronchitis, emphysema, active pulmonary tuberculosis, pulmonary carcinoma, pulmonary fibrosis, or pulmonary hypertension.
9. Have obstructive sleep apnea severe enough to warrant a prescription for biphasic or continuous positive-airway pressure therapy (BiPAP or CPAP), regardless of subject compliance with this therapy.
10. Taking any of the following medications:

    * Oral or parenteral beta blockers (excluding eye drops)
    * Strong cytochrome P450 3A4 inhibitors
    * Anti-IgE therapy, Xolair (omalizumab)
    * Monoamine oxidase (MAO) Inhibitors
    * Monoclonal antibodies/biologic agents which may affect the course of asthma (such as mepolizumab, reslizumab, lebrizumab, and others)
11. Had a viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks before Screening (Visit 1), or have such an infection during the Run-in Period.
12. Participated in an interventional study or used any investigational drug for any disease within 30 days (or 5 half-lives, if this is longer than 30 days) before Visit 1, or participated in this interventional study under the current protocol at any time previously.
13. Are hypersensitive to any β2-agonist sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy or any component of these combination medications including severe milk protein hypersensitivity.
14. Are exhibiting any factors (e.g., infirmity, disability, or geographic location, inability to follow instructions or study compliance requirements) that the investigator believes would likely limit the subject's compliance with the study protocol or scheduled site visits.
15. Have an affiliation with the participating site; in other words, subject may not be an immediate family member of any study site staff and may not be employed directly or indirectly by the study site.
16. Have a positive urine drug screen at Screening Visit.
17. Have a positive urine cotinine screen at Screening Visit.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1556 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
FEV1-time curve (day 1) | 24 hours
  Baseline-adjusted area under the serial FEV1-time curve calculated from time 0 (zero) to 12 hours on the first day of the Treatment Period
FEV1-time curve (day 28) | 24 hours
  Baseline-adjusted, pre-dose FEV1 on the last day of the Treatment Period

CONTACTS AND LOCATIONS:
Locations (1):
- West-Ward Research Site #1, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No